CLINICAL TRIAL: NCT02811055
Title: Pilot Study of Aprepitant Effect on Aldosterone Secretion in Diabetic Patient (Diabetes Mellitus) With Hypertension Associated With Low Renin
Acronym: APHOS-02
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2013/142/HP
Record Dates: First submitted 2016-05-25; First posted 2016-06-23 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Type 2 Diabetes; Hypertension
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension | interventions — Blood Specimen Collection; Electrocardiography

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Administration of Aprepitant (Experimental): Administration of Aprepitant 80 mg once per day during 14 days; Blood sampling, electrocardiogram, orthostatic test and Blood Pressure Measurement are done after 14 days
  Interventions: Biological: Blood sampling; Procedure: Blood Pressure Measurement; Device: electrocardiogram; Procedure: orthostatic test; Drug: Administration of Aprepitant
- Administration of placebo (Placebo Comparator): Administration of Placebo once per day during 14 days; Blood sampling, electrocardiogram, orthostatic test and Blood Pressure Measurement are done after 14 days
  Interventions: Biological: Blood sampling; Procedure: Blood Pressure Measurement; Device: electrocardiogram; Procedure: orthostatic test; Drug: Administration of placebo

INTERVENTIONS:
Biological: Blood sampling — Blood sampling for Plasma aldosterone, Plasma cortisol, plasma renin, plasma electrolytes after before and after administration of Aprepitant 80 mg once per day during 14 days or Administration of placebo once per day during 14 days
Procedure: Blood Pressure Measurement — Blood Pressure Measurement before and after Administration of Aprepitant 80 mg once per day during 14 days or administration of placebo once per day during 14 days
Device: electrocardiogram — Electrocardiogram before and after Administration of Aprepitant 80 mg once per day during 14 days or administration of placebo once per day during 14 days
Procedure: orthostatic test — Orthostatic test after Administration of Aprepitant 80 mg once per day during 14 days or administration of placebo once per day during 14 days
Drug: Administration of Aprepitant — Administration of Aprepitant 80 mg once per day during 14 days
  Arms: Administration of Aprepitant
Drug: Administration of placebo — Administration of placebo once per day during 14 days
  Arms: Administration of placebo

SUMMARY:
Aldosterone regulation is mediated by hormonal control, and nervous control. Autonomic nervous system action could be mediated by neuropeptides in the adrenal gland. Therefore, in pathological conditions and especially in diabetes, low-renin hypertension with normal or high plasma aldosterone could be caused by sympathetic nervous system hypertonia.

Data from the literature and previous in vitro research conducted in the investigators' laboratory (INSERM U982, University of Rouen) suggest that adrenal corticosteroid secretion might be controlled by sympathetic nervous system. This neurocrine regulation of corticosteroid secretion involves locally released neuropeptides. Among them, substance P is able to stimulate aldosterone and cortisol production via NK1 receptors. A previous clinical trial conducted at the University Hospital of Rouen, APHOS (NCT00977223) studied the effects of a NK1 receptor antagonist, aprepitant, on adrenocortical secretions in healthy volunteers.

The aim of the present study is to investigate the effects of a NK1 receptor antagonist, aprepitant, on adrenocortical secretions in volunteers with diabetes associated with low-renin hypertension. Aprepitant is a drug already available for the treatment of nausea induced by chemotherapy.

In the present phase II trial, plasma aldosterone and cortisol levels will be measured under treatment with aprepitant versus placebo, in both basal conditions and after activation of the adrenocortical function by upright posture. All volunteers will be given the two substances (aprepitant and placebo) in a random order during two 14 day-periods separated by a 21 day-wash-out.

This study should allow to determine the role of substance P in the control of corticosteroid production in human with diabetes, associated with a low-renin hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Male or menopausal female subjects;
* Age ranging 18-30 years old;
* Submitted to a social security regimen;
* Agreeing to the study & Informed consent form signed;
* Body mass index ([weight (kg)/height (m)]²) < 27;
* No treatment received 6 weeks before inclusion;
* No anomaly after: complete clinical examination, pulse and blood pressure measurement, ECG;
* No biological abnormality after the following biological testing:

Hematology: white & red blood cells & platelets count, haemoglobin, hematocrit, Blood biochemistry: sodium, potassium, chloride, bicarbonate, creatinine, urea, Urinary biochemistry (24 h collection): cortisol, aldosterone, Serologies: HIV, HBV, HCV,

* No participation in a clinical trial 3 months ago before inclusion,
* Subscription to national social security,
* Signed informed consent.

Exclusion Criteria:

* Female subject potentially pregnant,
* Subject younger than 18 year-old and older than 70 year-old,
* Subject without diabetes condition or with diabetes but normal blood pressure (below 130/80 mmHg),
* Subject with glycated hemoglobin HbA1c < 6.5% or >11%,
* Subject with leuconeutropenia (neutrophils below 1700/mm3),
* Subject with severe medical or surgical history,
* Patients treated with drugs metabolized by CYP3A4 and CYP2C9: corticosteroids, vitamin K , hormonal contraceptives, tolbutamide, benzodiazepines, derived from ergot, antiepileptics, hypericum, macrolides, azole antifungals.
* Patients treated with drugs interfering with the renin-angiotensin- aldosterone system : beta-blockers, diuretics , anti -aldosterone drugs , direct renin inhibitors , insulin,
* type 2 diabetes patients with a vegetative autonomic neuropathy,
* Patients with adrenal mass was diagnosed at imaging,
* hepatic or renal impairment (defined respectively by secondary clinical and biological manifestations altered hepatocyte functions or estimated glomerular filtration rate less than 60 mL / min / 1.73 m2);nephrotic syndrome (defined by hypoalbuminemia less than 30 g / L associated with proteinuria at 3 grams / 24 hours);edematous syndrome (defined by the presence of edema of the lower limbs),
* Orthostatic hypotension (defined by a decrease in systolic blood pressure of 20 mmHg and at least the diastolic blood pressure of 10 mmHg or more),
* arrhythmias or cardiac conduction,
* heart failure (NYHA class II minimum),
* epilepsy,
* serious psychiatric condition,
* Severe allergic history, hypersensitivity to aprepitant,
* People with hereditary problems of fructose intolerance, glucose malabsorption, galactose, or sucrase-isomaltase,
* People with lactose intolerance,
* subject unwilling or cannot be followed regularly. Persons deprived of their liberty by a judicial or administrative decision, those hospitalized without consent and those admitted to a health or social establishment for purposes other than research, the adults subject to a measure of legal protection or unable to consent may not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-07-13 (Actual); Primary Completion 2020-12-05 (Actual); Study Completion 2020-12-05 (Actual)

PRIMARY OUTCOMES:
Difference from baseline in Plasma aldosterone concentration | Baseline and Day 14
  Plasma aldosterone concentration is analyzed

SECONDARY OUTCOMES:
Difference from baseline in Plasma cortisol | Baseline and Day 14
  Plasma cortisol concentration is analyzed
Difference from baseline in plasma renin | Baseline and Day 14
  plasma renin concentration is analyzed
Difference from baseline in blood electrolytes measurement | Baseline and Day 14
  blood electrolytes concentration is analyzed
Difference from baseline in HOMA index | Baseline and Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Gaétan PREVOST, MD, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: No